CLINICAL TRIAL: NCT06926738
Title: Effect of Upper Thoracic Spine Manipulation on Cervical Symptoms and Selected Muscle Activities in Chronic Mechanical Neck Pain
Brief Title: Effect of Upper Thoracic Manipulation on Neck Pain and Selected Muscle Activities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Nagy Hassan Abdelhamid, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Upper thoracic manipulation
Record Dates: First submitted 2025-04-05; First posted 2025-04-15 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-01

CONDITIONS: Chronic Neck Pain
Keywords: Neck Pain; Thoracic manipulation; Manual Therapy; Neck pain with Mobility Deficits; Muscle activity
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upper thoracic manipulation group (Experimental): The Patients in this group will receive Upper Thoracic Manipulation.
  Interventions: Other: Upper Thoracic Manipulation
- Sham Upper Thoracic Manipulation (Sham Comparator): The patients in this group will receive the sham upper thoracic manipulation.
  Interventions: Other: Sham Comparison

INTERVENTIONS:
Other: Upper Thoracic Manipulation — Segmental mobility will be assessed using posteroanterior central vertebral pressure and posteroanterior unilateral vertebral pressure. It will be done while the patient lies in a prone position and the examiner stands at the level of the patient's head.
  Afterwards, the subjects in the thoracic manipulation group will be asked to lie in a prone position on a standard examination table and they were marked on both sides of the zygapophyseal joint of the selected segments including levels from T1- T4. Subjects will then be instructed to perform deep inhalation and exhalation and at the end of exhalation, the Clinician will perform thoracic manipulation (screw thrust technique) at the selected segmental level/s. This maneuver will be repeated for a maximum of two attempts in case of no hearing of a pop sound. It will be performed by an experienced physiotherapist with more than 10-year experience.
  Arms: Upper thoracic manipulation group
Other: Sham Comparison — Segmental mobility will be assessed using posteroanterior central vertebral pressure and posteroanterior unilateral vertebral pressure. It will be done while the patient lies in a prone position and the examiner stands at the level of the patient's head.
  Afterwards, the subjects in the thoracic manipulation group will be asked to lie in a prone position on a standard examination table and they were marked on both sides of the zygapophyseal joint of the selected segments including levels from T1- T4. Subjects will then be instructed to perform deep inhalation and exhalation and at the end of exhalation, the Clinician will just the place the hands on the selected levels in the same hand placement of Thoracic manipulation group (screw thrust technique) without applying the manipulation. It will be performed by an experienced physiotherapist with more than 10-year experience.
  Arms: Sham Upper Thoracic Manipulation

SUMMARY:
This study will investigate the immediate and short-term effects of upper thoracic manipulation versus sham upper thoracic manipulation on Pain intensity, Cervical ROM, the myoelectric activity of the sternocleidomastoid muscle and upper trapezius muscle during Maximum voluntary isometric contraction.

DETAILED DESCRIPTION:
This study will investigate the immediate and short-term effects of upper thoracic manipulation versus sham upper thoracic manipulation on Pain intensity measured by the visual analogue scale, Cervical ROM measured by CROM, the myoelectric activity of the sternocleidomastoid muscle and upper trapezius muscle during Maximum voluntary isometric contraction measured by Neuro-Soft using surface electrodes. All outcomes will be measured Pre-intervention, Immediately Post-Intervention, One-week Post-intervention, Two-week post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects diagnosed and classified as having chronic non-specific NP with mobility disorders based on clinical guidelines of NP:

   * Having NP for at least 3 months that may be associated with referred shoulder or upper extremity pain (Blanpied et al., 2017; Erdem et al., 2021; Puntumetakul et al., 2015).
   * Present with a limitation of cervical ROM and their pain can be provoked by sustained end-range spinal movements or positions will be included (Blanpied et al., 2017).
   * Patients present with unilateral or bilateral symptoms will be included (Blanpied et al., 2017; Yang et al., 2015).
2. Age between 18-40 (J. Dunning & Rushton, 2009)
3. Negative four tests of the Wainner cluster to exclude NP with radiating pain (Wainner et al., 2003).
4. Hypomobility of at least one of the upper thoracic vertebrae (T1-T4) during segmental mobility assessment (Ssavedra-Hernández et al., 2011).

Exclusion Criteria:

1. Subjects diagnosed as cervical radiculopathy or myelopathy (Ssavedra-Hernández et al., 2011).
2. A history of whiplash injury, past cervical or thoracic surgery, rheumatoid arthritis, spinal fracture, heart disease, a recent significant trauma, and meningitis (Joshi et al., 2020; Puntumetakul et al., 2015).
3. The presence of contraindications of spinal manipulation as spinal infection and spinal osteoporosis(Ssavedra-Hernández et al., 2011).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Pre-intervention, Immediately Post-Intervention, One-week Post-intervention, Two-week post-intervention.
  A hard copy of the Visual analogue scale will be given to the patient who will be asked to mark a perpendicular line between the two borders of the scale to express his/her pain level.
  It will be measured pre-treatment, post-treatment, and each week for 2 weeks. The level of pain will be measured at the end range of active extension.

SECONDARY OUTCOMES:
Cervical Range of Motion | Pre-intervention, Immediately Post-Intervention, One-week Post-intervention, Two-week post-intervention.
  The cervical ROM measurements will be performed with the participants sitting on a chair with instructions to sit in an upright posture. Prior to starting measurement, the patient will be asked to do these movements 5 times in each direction for familiarization and as a warm-up.
  The participant will sit erect with the thoracic spine away from the back of the chair, arms hanging at the sides, and feet flat on the floor. The participants were instructed to stare at a spot marked on a wall in front of them.
  Flexion, Extension, right and left side bending and rotation will be measured. Each measurement will be repeated for total three times.
Sternocleidomastoid muscle activity | Pre-intervention, Immediately Post-Intervention, One-week Post-intervention, Two-week post-intervention.
  Regarding EMG measurement of the sternocleidomastoid, the electrodes will be positioned over the sternocleidomastoid muscle at half the distance between the mastoid process of the temporal bone and the jugular notch of the sternum, slightly posterior to the center of the belly of the muscle, and parallel to the muscle fibers. The reference electrode will be attached to the proximal portion of the sternum with tape.
  Each participant will perform three 5-s MVIC for each muscle. Each subject will be asked to increase the force against the assessor's hand, reach the maximum effort, and hold it for EMG recording. The mean value of the three trials for the maximal contraction in each muscle will be taken.
  The patient will be supine lying and fully rested for the measurement of the SCM activity. To measure the MVIC of the Sternocleidomastoid muscle, the patient will be asked to flex the cervical spine against maximal resistance from the examiner on the forehead area while supine lying
Upper trapezius muscle activity | Pre-intervention, Immediately Post-Intervention, One-week Post-intervention, Two-week post-intervention.
  The Patient will be sitting in a chair with erect posture, hands supported on the thighs, feet parallel and supported on the floor, and eyes open for measurement of the upper trapezius muscle activity. The active and the reference electrodes will be placed 2 cm lateral to the midpoint between C7 and posterior acromion with 2 cm inter-electrode distance and ground placed on C7.
  Each participant will perform three 5-s MVIC for each muscle. Each subject will be asked to increase the force against the assessor's hand, reach the maximum effort, and hold it for EMG recording. The mean value of the three trials for the maximal contraction in each muscle was taken as the MVIC. The rest time between each maximum contraction will be 30 seconds. To measure the MVIC of the upper trapezius muscle, the patient will be asked to abduct his/her shoulder to 90 degrees with the elbow fully extended against maximum resistance which will be applied superior to the elbow to resist abduction.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - CairoU, Giza
  - Faculty of Physical Therapy, Cairo University, Giza

IPD SHARING:
Plan to Share IPD: No